CLINICAL TRIAL: NCT05879770
Title: Is the Use of Prolene as Sufficient as the Use of Wire in Shouldice Surgery to Keep the Recurrence Rate Low After One Year?
Acronym: Wire vs Prolen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shouldice Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: #2023-02
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Inguinal Hernia
Keywords: Hernia, Shouldice Repair, groin hernia
MeSH Terms: conditions — Hernia, Inguinal; Hernia | interventions — Sutures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wire group: Patients who underwent Shouldice inguinal hernia repair using wire.
  Interventions: Other: suture material
- prolene group: Patients who underwent Shouldice inguinal hernia repair using prolene.
  Interventions: Other: suture material

INTERVENTIONS:
Other: suture material — Some patients have had a shouldice repair with wire in the past and others with Prolene.

SUMMARY:
When conducting the Shouldice procedure the 4-layer suture of the transversalis fascia is usually done with Prolene worldwide. At the Shouldice hospital the wire has originally been used for these augmentation. During the last decade several Shouldice Surgeons started to use the Prolene due to occasional delivery problems of the wire from Germany.

The 1-year- recurrence rate at the Shouldice hospital is 1,15% (mainly wire-use). The published 1-year recurrence rate in Europe is 2%.

As quality assessment, this project intends to evaluate these two options for suturing (wire vs Prolene) in the elective inguinal hernia patient in terms of 1-year recurrence rate. The population of focus will be those who had a primary or secondary inguinal hernia operation at Shouldice Hospital and the project is estimated to take 3 months.

DETAILED DESCRIPTION:
a. Study design A total of 1400 patients (n=700 with wire; n=700 with Prolene) who underwent Shouldice surgery at Shouldice Hospital will be contacted by telephone. They will be asked whether a relapse occurred after their surgery.

Sample size calculation:

The 1-year recurrence rate at Shouldice Hospital is 1.15% (mainly wire use). The published 1-year recurrence rate in Europe is 2% [1-3]. Statistics: non-inferiority: delta for non-inferiority (defined equivalence range) = 1%. Total N = 1120 (0% dropout), with 20% dropout: N = 1400.) The same number of patients will be analyzed with regard to Shouldice repair due to a first relapse (time period of data extraction 2019-2021).

Since over 6000 hernias are operated annually, a consecutive data extraction of patients operated in 2021 will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of all sexes who have undergone inguinal hernia surgery in Shouldice technique.

Exclusion Criteria:

* Hernia repair using a mesh

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients of all sexes who have undergone inguinal hernia surgery in Shouldice technique.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 1 year
  One-year recurrence rate

SECONDARY OUTCOMES:
Reoperation rate due to a recurrence | 1 year
  Reoperation rate due to a recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Shouldice Hospital, Thornhill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided